CLINICAL TRIAL: NCT07343336
Title: FENUA-METABOGOUT : Genetic Landscape of Gout, Inflammation and Metabolic Diseases in French Polynesia.
Brief Title: Landscape of Gout in French Polynesia.
Acronym: METABOGOUT
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Variant Bio, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC-P00126
Record Dates: First submitted 2025-10-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gout Disease; Metabolic Diseases; Inflammation
Keywords: Gout disease; metabolic disease; inflammation
MeSH Terms: conditions — Metabolic Diseases; Inflammation | interventions — Epidemiologic Studies; Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample, urine sample, synovial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General Population Group: Patients aged between 18 and 75 years old who did not take part in the TOPATA study in 2021 and who visit their general practitioner for a consultation (for whatever reason)
  Interventions: Other: Epidemiological study; Diagnostic Test: Blood and urine tests
- Gout Group: Patients aged between 18 and 75 years old who are treated at the rheumatology clinic of the Taaone Hospital Centre (CHT) in Papeete by Dr Baptiste Gérard.
  * There is a tophaceous gout subgroup: patients with tophaceous gout.
  * And a gout attack subgroup: patients presenting with a gout crisis.
  Interventions: Other: Epidemiological study; Diagnostic Test: Blood and urine tests
- Follow-up group 2021: Patients aged between 18 and 75 years old who were included in the TOPATA study in 2021 and for whom genetic and biological samples during the 2021 study were taken.
  Patients must have had hyperuricaemia without signs of gout OR without hyperuricaemia or gout at the time of inclusion in the 2021 TOPATA study.
  Interventions: Other: Epidemiological study; Diagnostic Test: Blood and urine tests

INTERVENTIONS:
Other: Epidemiological study — Collection of sociodemographic data, collection of treatment data, standard and clinical ophthalmological examination, physical and biological measurements, clinical characteristics specific to chronic and metabolic diseases, questionnaires (gout questionnaire, health assessment questionnaire (HAQ-II), EuroQol (EQ)-5D-5L, joint pain, state of health, diet and physical activity, access to care, addictions, sleep quality, pain scale (EVA), personal and family history) will be performed.
Diagnostic Test: Blood and urine tests — Collection of blood and urine samples for genetic, biochemical, omics, and biobank analyses, in order to characterize cardiometabolic health markers will be performed.

SUMMARY:
The aim of this research is to characterise the genetic and molecular landscape of gout, inflammation and metabolic diseases, as well as the associated molecular, anthropomorphic and pathological characteristics.

DETAILED DESCRIPTION:
Recent work by the GHICL has highlighted the imminent public health problem represented by gout and hyperuricaemia in French Polynesia, with gout affecting around 15% and hyperuricaemia 71.6% of the adult population.

Hyperuricaemia is defined as a serum urate level above the saturation point, leading to its crystallisation under biological conditions. It is generally accepted that hyperuricaemia (HU) begins at 6.0 mg/dL (360 µmol/L).

The best-known consequence of hyperuricaemia is the development of gout, which results from the inflammatory response to the presence of monosodium urate (MSU) crystals in and around the joints. The factors modulating the deposition of MSU crystals in HU are poorly understood and a potential genetic contribution is unknown. It is known that the inflammatory response to the presence of MSU crystal deposits causing gout flares is mediated by activation of the NLRP33 inflammasome, but there is significant variability in this inflammatory response within the same individual (irregular recurrence of flares), and between individuals. The exceptionally high prevalence of HU that have been identified in French Polynesia represents a major health burden, as hyperuricaemia and gout are associated with many other cardiometabolic diseases.

For example, hyperuricaemia, BMI and type 2 diabetes are all associated with the risk of gout. The association between gout and cardiovascular events is also well known, and is thought to be mediated by a persistent inflammatory state. These data are particularly relevant in the context of French Polynesia where, in addition to high rates of gout and HU, a prevalence of obesity of over 40% (BMI >30kg/m2) and a prevalence of diabetes (based on HBA1c measurements) of over 13% was previously identified by the same team.

This last point is particularly striking as the prevalence of diabetes based on self-reported diagnosis was only 7%, indicating that many people are probably undiagnosed and therefore untreated. A better understanding not only of the mechanism and causal link between these conditions and risk factors, but also of the genetic basis of the disease, could lead to the development of therapies and to the improvement in diagnosis. This is particularly crucial in French Polynesia, where hyperuricaemia and its pathological effects on cardiometabolic health affect a large proportion of the adult population.

Here a multi-pronged approach to take advantage of a previous study named 'TOPATA' (NCT04812886) performed previously in French Polynesia, is proposed. The idea is to expand the existing cohort, in order to identify the genetic effectors contributing to the high rates of metabolic diseases previously observed, and to track the longitudinal impacts of HU.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Age between 18 and 75 years old inclusive
* Signature of informed consent
* Fasting for the collection of biological samples
* Declared Polynesian ancestry
* Affiliated to a social security scheme

General population group :

* Not having participated to the 2021 TOPATA study
* Visiting a general practitioner (for whatever reason)

Gout Group :

* Managed at the rheumatology clinic of the Taaone Hospital Centre (CHT) in Papeete by Dr Baptiste Gérard.

Tophaceous gout sub-group:

* Present with tophaceous gout.

Gout crisis subgroup:

* Be within 48 hours of the onset of a gout attack
* Agree to return 1 week after inclusion for the second blood and urine sample.

  2021 follow-up group:
* To have been included in the TOPATA study in 2021
* Have taken the genetic and biological samples that generated the genetic and serum urate data for the 2021 study
* Have hyperuricaemia without signs of gout OR without hyperuricaemia or gout at the time of inclusion in TOPATA

Exclusion Criteria:

All participants :

* Refusal or inability to understand or give consent
* Physical inability to follow and respect the protocol
* 1st degree relative*,
* Person under guardianship or trusteeship
* Pregnant or breast-feeding woman

  * If several relatives from the same household are eligible to participate, only one person may be included in the study. The choice is left to the discretion of the investigator or the first person met. However, both members of a couple (e.g. husband and wife) may participate.
* General population group :
* Unable to return for sampling if required.
* Gout group :
* Person wearing a knee prosthesis
* People suffering from other inflammatory rheumatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population group: Participants will be recruited by general practitioners or study nurses during consultations in community-based practices. The objective is to include a representative general population sample, with no specific reason for consultation required or excluded.
  Gout group: Patients will be recruited at the Rheumatology Clinic of the Taaone Hospital Center (CHT) in Papeete when presenting with gout symptoms, either tophaceous gout or an acute flare within the previous 48 hours.
  2021 follow-up group: Participants from the TOPATA study conducted in 2021 will be recontacted by telephone to assess willingness to participate, followed by an in-person inclusion visit. Only individuals currently living in Tahiti will be contacted. Nurses will be responsible for recruitment, biological sample collection, physical measurements, and questionnaire administration.
Sampling Method: Non-Probability Sample
Enrollment: 2750 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
GWAS-identified associations between population-enriched genetic variants and health-related traits | 12 month
  Effect estimates (odds ratios or beta coefficients) for statistically significant associations between population-enriched genetic variants and predefined health-related traits identified through GWAS.

SECONDARY OUTCOMES:
Multiple correlation between gout, hyperuricemia, type 2 diabetes and obesity | 12 month
  Anthropometric and biological characteristics of gout, hyperuricemia, type 2 diabetes, and obesity will be assessed, and comorbidity associations analyzed using multivariate logistic regression. Measurements will include waist and hip circumferences, blood pressure, muscle properties by myotonometry, lower-limb strength via chair stand test, and handgrip strength. Blood analyses will assess lipid profile, liver function, inflammation, renal function and metabolism, glucose metabolism, and complete blood count. Urine analyses will also be performed.
Incidence rate of gout or HU in French Polynesia between 2021 and 2025 | 4 years
  Incidence rate of gout or HU in French Polynesia between 2021 and 2025 in a sample of participants in the 2021 cohort with asymptomatic HU and no gout.
Proportion of each type of urate-lowering therapy prescribed annually between 2019 and 2025 | 4 years
  Breakdown of types of THU prescribed between 2019 and 2025 based on the database of healthcare claims submitted to the Caisse de Prévoyance Sociale (CPS)
Incidence of major adverse cardiovascular events (MACE) in patients with gout, diabetes, or obesity | 12 month
  Occurrence of MACE related to gout, diabetes or obesity on the Healthcare Claims Database (HCD).
Determinants of progression from asymptomatic hyperuricemia (in 2021) to gout (in 2025) | 4 years
  Factors influencing the transition from asymptomatic HU to gout will be sought among demographic, anthropomorphic and biological characteristics, comorbidities, current treatments, genetic profiles, gene expression, proteomic profiles and metabolomic profiles.
Multiple correlation between metabolic changes and disease evolution | 12 month
  Severe gout is defined by subcutaneous tophi. Clinical characteristics will be assessed, including disease features (age at onset, duration), topography (affected joints, mono-/polyarticular and axial involvement), number, duration, and severity of flares, serum uric acid, and presence, number, and size of tophi. Treatment history and response (urate-lowering therapy, flare management), comorbidities (cardiovascular disease, chronic kidney disease, metabolic syndrome, diabetes, obesity, hypertension), and lifestyle factors (diet, alcohol, physical activity) will also be recorded. Molecular and biological characterization will include genetic, transcriptomic, proteomic, and metabolomic analyses to identify biomarkers associated with disease severity and progression.
Multiple correlation between molecular, clinical features and gout severity | 12 month
  Severe gout is defined by subcutaneous tophi. Clinical characteristics will be evaluated, including disease features (age at onset, duration), topography (affected joints, mono-/polyarticular and axial involvement), number, duration, and severity of flares, serum uric acid, and presence, number, and size of tophi. Treatment history and response (urate-lowering therapy, flare management), comorbidities (cardiovascular disease, chronic kidney disease, metabolic syndrome, diabetes, obesity, hypertension), and lifestyle factors (diet, alcohol, physical activity) will also be recorded. Molecular and biological characterization will include genetic, transcriptomic, proteomic, and metabolomic analyses to identify biomarkers linked to disease severity and progression.
Multiple correlation between gout attacks, clinical manifestations, gene expression, proteomic, and metabolomic profiles. | 12 month
  Gout attack characteristics will be investigated, including attack location (affected joints, mono- or polyarticular), pain intensity (VAS or NRS), and inflammatory parameters (CRP, ESR if available, leukocyte count and differential). Synovial fluid analysis will include total and differential cell counts and presence of monosodium urate crystals. Triggering factors (diet, alcohol, trauma, infection, medications), associated acute conditions (infection, surgery, cardiovascular events), and flare duration and severity will be recorded. Treatments and clinical response will also be documented. Molecular characterization will include genetic analyses (urate transport and inflammation variants), gene expression, proteomic profiling of blood and synovial fluid, and metabolomic analyses of serum, urine, and synovial fluid to identify biomarkers of acute flares.
Change in clinical and molecular characteristics of acute gout flares between baseline and 1-week visit | one week
  Composite assessment of acute gout flares including clinical characteristics (attack location, mono- or polyarticular involvement, pain intensity measured by VAS or NRS, inflammatory markers [CRP, ESR if available, leukocyte count and differential]), synovial fluid findings (total and differential cell counts and presence of monosodium urate crystals), triggering factors and associated acute conditions, flare duration and severity, treatments administered and clinical response, and molecular biomarkers identified through genetic analyses, gene expression profiling, proteomic analyses, and metabolomic profiling of blood, urine, and synovial fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, Professor, Principal Investigator — GHICL
Locations (6):
- French Polynesia (6):
  - Medical Office Dr Antoine Scuiller, Faa'a
  - Medical Office Dr Cedric Gueguen, Papeete
  - Medical Office Dr Voradeth Nouanesengsy, Papeete
  - CH de Polynesie Française Papeete, Pirae
  - Medical Office Dr Nanethida Nouanesengsy, Pirae
  - Medical Office Dr Raphael Habib, Pirae

IPD SHARING:
Plan to Share IPD: No